CLINICAL TRIAL: NCT04979949
Title: Double-Blind, Randomized, Controlled, Multi-Centered, Phase 2 Clinical Trial to Determine the Safety, Efficacy, and Immunogenicity of Booster Vaccination Against SARS-CoV-2
Brief Title: Booster Vaccination Against COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Hibrid COV-Rapel TR
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Sars-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 Vaccine; Booster; Efficacy; Immunogenicity; Safety
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; TURKOVAC

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Controlled, Multi-Center Phase 2 Clinical Trial to Determine Safety, Efficacy, and Immunogenicity of Booster Vaccination Against SARS-CoV-2 (Hybrid COV-Rapel TR)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CoronaVac (Active Comparator): Inactivated SARS-CoV-2 virus antigen, single intramuscular injection for boosting dose.
  Interventions: Biological: CoronaVac
- Turkovac (Experimental): Inactivated SARS-CoV-2 virus antigen, single intramuscular injection for boosting dose.
  Interventions: Biological: Turkovac

INTERVENTIONS:
Biological: CoronaVac — One dose vaccine will be administered to subjects who have passed at least 90 days and at most 270 days after the second dose of the first course of CoronaVac vaccine.
  Arms: CoronaVac
Biological: Turkovac — One dose vaccine will be administered to subjects who have passed at least 90 days and at most 270 days after the second dose of the first course of CoronaVac vaccine.
  Arms: Turkovac

SUMMARY:
A booster dose of vaccine (Turkovac or CoronaVac) will be administered to subjects who have passed at least 90 days and at most 270 days after the second dose of the first course of CoronaVac vaccine.

DETAILED DESCRIPTION:
To determine the safety and immunogenicity of booster doses of vaccine against SARS-CoV2 after a minimum of 90 days and a maximum of 270 days after the 2nd dose of a homologous 2 dose primary regimen.

It is planned to recruit 111 subjects for 2 vaccines (Turkovac and CoronaVac). There will be a total of 222 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy male or female aged 18 - 60 years (including both groups)
* Subjects who were vaccinated with CoronaVac for 2 doses and who had a minimum of 90 days and a maximum of 270 days after the second dose
* Subjects may have a controlled or moderate comorbidity
* Female subjects of childbearing potential should be willing to ensure that they or their partner use effective birth control methods continuously from 1 month before and up to 3 months after vaccination
* Subjects agreed to comply with all study requirements
* Subjects are willing to share their medical history with their physician and allow access to all medical records when relevant to study procedures
* Subjects are willing to agree to abstain from donating blood during the study

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

* Administration of any vaccine (registered or investigational) other than study intervention within 30 days before and after each study vaccine (one week for authorized seasonal flu vaccine or pneumococcal vaccine)
* Positive for COVID-19 after primary vaccination
* Pre-or planned use of another vaccine or product likely to affect the study (e.g. adenovirus vectored vaccines, any coronavirus vaccine)
* Subjects who were pregnant at the time of enrollment or who plan to become pregnant within the first 3 months following vaccination and who are breastfeeding
* Subjects with fever (above 38°C) at the time of vaccination and/or up to 72 hours before
* Administration of immunoglobulins and/or any blood product within 3 months prior to vaccination
* Any confirmed or suspected immunosuppressive or immunodeficiency state; asplenia; recurrent severe infections and use of immunosuppressants (less than ≤14 days) in the last 6 months, excluding topical steroids or short-term oral steroids
* Possible history of allergic disease or reaction (e.g. to the active substance) by any component of the study vaccines
* Any history of anaphylaxis
* Current cancer diagnosis or treatment (excluding basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venipuncture
* Continued use of anticoagulants such as coumarins and related anticoagulants (i.e. warfarin) or new oral anticoagulants (i.e. apixaban, rivaroxaban, dabigatran and edoxaban)
* Cerebral venous sinus thrombosis, antiphospholipid syndrome, or a history of heparin-induced thrombocytopenia and thrombosis (HITT or HIT type 2).
* Suspected or known current alcohol or drug addiction
* Any other significant disease, disorder or finding that could significantly increase the subject's risk for participation in the study, affect the subject's ability to participate in the study, or impair the interpretation of study data; severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, kidney disease, endocrine disorder, and neurological disease (mild/moderate well-controlled comorbidities are permitted)
* History of active or previous autoimmune neurological disorders (e.g. multiple sclerosis, Guillain-Barre syndrome, transverse myelitis) (Bell's palsy will not be an exclusion criterion)
* Subjects with severe renal impairment or liver failure
* Subjects who will undergo scheduled elective surgery during the study
* Subjects with a life expectancy of less than 6 months
* Subject who participated in another clinical trial study involving an investigational product in the past 12 weeks
* In case of clinical necessity, a COVID-19 PCR (polymerase chain reaction) test will be requested from the subjects, and subjects who are positive will be excluded from the study
* Known history of SARS-CoV-2 infection
* Acute respiratory disease (moderate or severe illness with or without fever) (Subjects may be screened again after acute condition has resolved)
* Fever (oral temperature > 37.8°C) (Subjects can be enrolled again after acute condition improves)
* Insufficient level of Turkish to perform the informed consent, except where briefing by an independent witness can be provided and is available

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 222 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 7 days after vaccination
  Incidence of adverse reactions within 7 days of vaccination in all subjects
Incidence of Serious Adverse Events (SAE) | 168 days after vaccination
  Incidence of Serious Adverse Events (SAE) in all subjects 168 days after vaccination

SECONDARY OUTCOMES:
Neutralizing antibody and anti-spike protein immunoglobulin G | On days 0, 28 and 84
  Amount of SARS-CoV2 anti-spike protein immunoglobulin G and SARS-CoV2 neutralizing antibody amount

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Omma, Assoc. Prof., Principal Investigator — Faculty Member
Locations (4):
- Turkey (Türkiye) (4):
  - Ankara City Hospital Internal Medicine Clinic, Ankara
  - Sancaktepe Martyr Professor Dr. İlhan Varank Training and Research Hospital Infectious Diseases and Clinical Microbiology Clinic, Istanbul
  - T.R. Ministry of Health Kartal Dr. Lütfi Kirdar City Hospital Infectious Diseases, Istanbul
  - Ümraniye Training and Research Hospital Infectious Diseases, Istanbul

REFERENCES:
- [Background] Kumar A, Singh R, Kaur J, Pandey S, Sharma V, Thakur L, Sati S, Mani S, Asthana S, Sharma TK, Chaudhuri S, Bhattacharyya S, Kumar N. Wuhan to World: The COVID-19 Pandemic. Front Cell Infect Microbiol. 2021 Mar 30;11:596201. doi: 10.3389/fcimb.2021.596201. eCollection 2021. PMID 33859951
- [Background] Dan JM, Mateus J, Kato Y, Hastie KM, Yu ED, Faliti CE, Grifoni A, Ramirez SI, Haupt S, Frazier A, Nakao C, Rayaprolu V, Rawlings SA, Peters B, Krammer F, Simon V, Saphire EO, Smith DM, Weiskopf D, Sette A, Crotty S. Immunological memory to SARS-CoV-2 assessed for up to 8 months after infection. Science. 2021 Feb 5;371(6529):eabf4063. doi: 10.1126/science.abf4063. Epub 2021 Jan 6. PMID 33408181
- [Background] Doria-Rose N, Suthar MS, Makowski M, O'Connell S, McDermott AB, Flach B, Ledgerwood JE, Mascola JR, Graham BS, Lin BC, O'Dell S, Schmidt SD, Widge AT, Edara VV, Anderson EJ, Lai L, Floyd K, Rouphael NG, Zarnitsyna V, Roberts PC, Makhene M, Buchanan W, Luke CJ, Beigel JH, Jackson LA, Neuzil KM, Bennett H, Leav B, Albert J, Kunwar P; mRNA-1273 Study Group. Antibody Persistence through 6 Months after the Second Dose of mRNA-1273 Vaccine for Covid-19. N Engl J Med. 2021 Jun 10;384(23):2259-2261. doi: 10.1056/NEJMc2103916. Epub 2021 Apr 6. No abstract available. PMID 33822494
- [Background] Wu K, Werner AP, Koch M, Choi A, Narayanan E, Stewart-Jones GBE, Colpitts T, Bennett H, Boyoglu-Barnum S, Shi W, Moliva JI, Sullivan NJ, Graham BS, Carfi A, Corbett KS, Seder RA, Edwards DK. Serum Neutralizing Activity Elicited by mRNA-1273 Vaccine. N Engl J Med. 2021 Apr 15;384(15):1468-1470. doi: 10.1056/NEJMc2102179. Epub 2021 Mar 17. No abstract available. PMID 33730471
- [Background] Madhi SA, Baillie V, Cutland CL, Voysey M, Koen AL, Fairlie L, Padayachee SD, Dheda K, Barnabas SL, Bhorat QE, Briner C, Kwatra G, Ahmed K, Aley P, Bhikha S, Bhiman JN, Bhorat AE, du Plessis J, Esmail A, Groenewald M, Horne E, Hwa SH, Jose A, Lambe T, Laubscher M, Malahleha M, Masenya M, Masilela M, McKenzie S, Molapo K, Moultrie A, Oelofse S, Patel F, Pillay S, Rhead S, Rodel H, Rossouw L, Taoushanis C, Tegally H, Thombrayil A, van Eck S, Wibmer CK, Durham NM, Kelly EJ, Villafana TL, Gilbert S, Pollard AJ, de Oliveira T, Moore PL, Sigal A, Izu A; NGS-SA Group; Wits-VIDA COVID Group. Efficacy of the ChAdOx1 nCoV-19 Covid-19 Vaccine against the B.1.351 Variant. N Engl J Med. 2021 May 20;384(20):1885-1898. doi: 10.1056/NEJMoa2102214. Epub 2021 Mar 16. PMID 33725432
- [Derived] Omma A, Batirel A, Aydin M, Yilmaz Karadag F, Erden A, Kucuksahin O, Armagan B, Guven SC, Karakas O, Gokdemir S, Altunal LN, Buber AA, Gemcioglu E, Zengin O, Inan O, Sahiner ES, Korukluoglu G, Sezer Z, Ozdarendeli A, Kara A, Ates I. Safety and immunogenicity of inactive vaccines as booster doses for COVID-19 in Turkiye: A randomized trial. Hum Vaccin Immunother. 2022 Nov 30;18(6):2122503. doi: 10.1080/21645515.2022.2122503. Epub 2022 Oct 31. PMID 36315843